CLINICAL TRIAL: NCT07167576
Title: Computer-based Tutorial as Supportive Means to Enhance Quality and Efficiency of the Informed Consent Process for Cataract Surgery:
Brief Title: Computer-based Tutorial as a Means to Enhance the Informed Consent Process for Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Purpose: Other
Other Study IDs: CAT
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2010-09

CONDITIONS: Patients' Information Level About Cataract Surgery; Patients' Attitude Before and After Cataract Surgery
MeSH Terms: interventions — Physicians

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Catinfo and discussion group (Active Comparator): Patients watch a short computer presentation on the Catinfo tool before the discussion with the physician
  Interventions: Other: Catinfo tool and discussion with physician
- Discussion group (Active Comparator): Patients have the standard discussion with the physician
  Interventions: Other: discussion with physician

INTERVENTIONS:
Other: Catinfo tool and discussion with physician — Patients in the study group watch a computer presentation with information about the cataract surgery
  Arms: Catinfo and discussion group
Other: discussion with physician — Patients in the control group have a discussion with the physician
  Arms: Discussion group

SUMMARY:
Informing the patient and obtaining the informed consent is one of the major duties physicians perform before beginning a medical treatment.

Some years ago we developed the so-called CatInfo programme that allows to inform the patient inter-actively prior to the face-to-face interview with the physician. This program was found to lead to significantly better informed patients in our hospital. Although these findings were significant, we would like to investigate more on two other aspects in this study: Firstly, we would like to learn more about the patients' attitude before and after surgery. Therefore, we would like to ask the patients' about their willingness of being informed and decision making using a standardised questionnaire. Secondly, we would like to investigate on the differences in the duration of informed consent taking in patients that have heard and seen the CatInfo vs. patients received no information prior to the face-to-face interview with the physician. Patients will be randomly assigned to one of these groups.

This difference will then be evaluated together with the result of the MCQ (assessing the patients' knowledge concerning cataract surgery after informed consent taking). The primary hypothesis is that patients' are better informed after watching the CatInfo tool although the face-to face interview is shorter.

DETAILED DESCRIPTION:
Informing the patient and obtaining the informed consent is one of the major duties physicians perform before beginning a medical treatment. At the same time expectations of patients in modern medicine grow and so do the legal requirements on informing the patient. Studies have shown that patients often cannot remember the most important and essential parts of the communication with their physician.

It also appears that the use of printed information sheets providing patient information has not really changed this situation.

By the law of many countries, the duty to inform the patient has to be carried out in a personal face-to face communication of patient and physician. Frequently, the informed consent of the patient is documented by signature on printed forms and only a brief discussion is performed. Additionally, due to the asymmetry in the relationship between patient and physician, patients will often hesitate to ask questions in case of poor understanding of either their diagnosis or the planned procedure. Therefore, the informed consent process may not be sufficient to satisfy the patient's needs.

All these factors can result in misunderstandings, poor comprehension of the planned procedure and dissatisfied patients and may eventually lead to litigation.

Some years ago we developed the so-called CatInfo programme that allows to inform the patient inter-actively prior to the face-to-face interview with the physician. This program was found to lead to significantly better informed patients in our hospital. Although these findings were significant, we would like to investigate more on two other aspects in this study: Firstly, we would like to learn more about the patients' attitude before and after surgery. Therefore, we would like to ask the patients' about their willingness of being informed and decision making using a standardised questionnaire. Secondly, we would like to investigate on the differences in the duration of informed consent taking in patients that have heard and seen the CatInfo vs. patients received no information prior to the face-to-face interview with the physician. This difference will then be evaluated together with the result of the Multiple choice questionnaire (assessing the patients' knowledge concerning cataract surgery after informed consent taking). The primary hypothesis is that patients' are better informed after watching the CatInfo tool although the face-to face interview is shorter.

Patients will be randomly allocated to the study or the control group. Additionally all patients will be called one month after surgery to assess their satisfaction with the informed consent process.

ELIGIBILITY:
Inclusion Criteria:

* Cataract
* Age 18 and older
* First eye to be operated
* No previous ophthalmic surgery
* written informed consent to participation in the study

Exclusion Criteria:

* Visual acuity of less than 0.1 Snellen in the worse eye
* Severe hearing loss
* Inability to use touch screen device (e.g. severe tremor, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
patients' attitude before and after cataract surgery | one month
  assessed by validated questionnaires

SECONDARY OUTCOMES:
- Difference concerning duration of the face to face interview with the physician between both groups | one hour
  measured in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Vienna, Austria